CLINICAL TRIAL: NCT06838650
Title: Beneficial Effects of Low-Dose Intravenous Dexmedetomidine Premedication in Patient Undergoing Laparoscopic Cholecystectomy Under General Anesthesia
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Atia Medhat Atia Bakhet, Residant doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LD Dex premedication LC
Record Dates: First submitted 2025-02-19; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Laparoscopic Cholecystectomy Surgery
Keywords: Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Placebo Comparator): patients undergoing laparoscobic cholestotectomy will be premedicated with saline . The patients will be premedicated before anesthesia induction
  Interventions: Drug: Saline
- Group B (Active Comparator): patients undergoing LC will be premedication with 0.5 µg/kg Dex. The patients will be premedicated before anesthesia induction
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — patients will recive of low-dose (0.5 µg/kg) intravenous Dexmedetomidine before general anathesia
  Arms: Group B
Drug: Saline — patients will recive saline
  Arms: Group A

SUMMARY:
Laparoscopic cholecystectomy (LC) is considered the standard treatment for gallbladder disease.1 Compared to open cholecystectomy, LC is the preferred treatment approach because it is associated with less surgical trauma, shorter hospital stays, and faster postoperative recovery.2 However, the elevated intra-abdominal pressure due to pneumoperitoneum can cause various stress responses that affect patient prognosis and present a severe challenge in anesthetic management.3 Therefore, the search for an optimal anesthetic protocol to minimize adverse reactions during LC remains critical.

Dexmedetomidine (Dex), a potent and highly selective α2-adrenergic receptor agonist, presents sedative, analgesic, anesthetic, and sympatholytic properties, without causing respiratory depression, when used in an appropriate dose range.4 Numerous studies have suggested that Dex can effectively attenuate the surgical stress response and provide intraoperative hemodynamic stability.5 Furthermore, it has been shown to reduce anesthetic requirements and improve the quality of patient recovery.6,7 Hence, it has been widely used as an adjuvant during general anesthesia.

Nevertheless, the clinical effects of Dex remain controversial. Some studies have shown that the anesthesia recovery time is prolonged and the incidence of bradycardia increases significantly after intravenous Dex infusion.8-10 This is mainly attributed to the different doses and methods of Dex administration. Although the complications are always transient and reversible, timely attention is required to avoid serious adverse consequences. To enhance the value of Dex for clinical application and improve the quality of general anesthesia, the more appropriate protocol of Dex administra- tion need to be explored. The elimination half-life of Dex is approximately 2 h, with a rapid distribution half-life of approximately 6 min.11 Most LC procedures are completed within 1 h; therefore, to reduce postoperative complications and shorten postoperative recovery time, we prefer preoperative Dex loading to intraoperative continuous Dex infusion. According to our previous data, the anesthesia awakening time will be prolonged and the incidence of bradycardia increased significantly when 1.0 µg/kg of Dex will be administered before general anesthesia induction. This prospective, double-blind, randomized controlled trial aimed to determine the efficacy of low-dose (0.5 µg/kg) intravenous Dex premedication on hemodynamics and adverse events during general anesthesia. We aimed to confirm the efficacy of low- dose intravenous Dex premedication in patients under general anesthesia during LC and to provide a data reference for the clinical application of Dex in further research. Dexmedetomidine (Dex) is a potent and highly selective α2-adrenergic receptor agonist. Within an appropriate dose range, Dex can effectively attenuate the surgical stress response, provide intraoperative hemodynamic stability, and improve the patient recovery quality. High-dose Dex can delay patient awakening from anesthesia and increase the incidence of bradycardia. This randomized controlled trial aimed to investigate the effects of low-dose intravenous Dex premedication in patients undergoing laparoscopic cholecystectomy (LC).

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy (LC) is considered the standard treatment for gallbladder disease.1 Compared to open cholecystectomy, LC is the preferred treatment approach because it is associated with less surgical trauma, shorter hospital stays, and faster postoperative recovery.2 However, the elevated intra-abdominal pressure due to pneumoperitoneum can cause various stress responses that affect patient prognosis and present a severe challenge in anesthetic management.3 Therefore, the search for an optimal anesthetic protocol to minimize adverse reactions during LC remains critical.

Dexmedetomidine (Dex), a potent and highly selective α2-adrenergic receptor agonist, presents sedative, analgesic, anesthetic, and sympatholytic properties, without causing respiratory depression, when used in an appropriate dose range.4 Numerous studies have suggested that Dex can effectively attenuate the surgical stress response and provide intraoperative hemodynamic stability.5 Furthermore, it has been shown to reduce anesthetic requirements and improve the quality of patient recovery.6,7 Hence, it has been widely used as an adjuvant during general anesthesia.

Nevertheless, the clinical effects of Dex remain controversial. Some studies have shown that the anesthesia recovery time is prolonged and the incidence of bradycardia increases significantly after intravenous Dex infusion.8-10 This is mainly attributed to the different doses and methods of Dex administration. Although the complications are always transient and reversible, timely attention is required to avoid serious adverse consequences. To enhance the value of Dex for clinical application and improve the quality of general anesthesia, the more appropriate protocol of Dex administra- tion need to be explored. The elimination half-life of Dex is approximately 2 h, with a rapid distribution half-life of approximately 6 min.11 Most LC procedures are completed within 1 h; therefore, to reduce postoperative complications and shorten postoperative recovery time, we prefer preoperative Dex loading to intraoperative continuous Dex infusion. According to our previous data, the anesthesia awakening time will be prolonged and the incidence of bradycardia increased significantly when 1.0 µg/kg of Dex will be administered before general anesthesia induction. This prospective, double-blind, randomized controlled trial aimed to determine the efficacy of low-dose (0.5 µg/kg) intravenous Dex premedication on hemodynamics and adverse events during general anesthesia. We aimed to confirm the efficacy of low- dose intravenous Dex premedication in patients under general anesthesia during LC and to provide a data reference for the clinical application of Dex in further research. Dexmedetomidine (Dex) is a potent and highly selective α2-adrenergic receptor agonist. Within an appropriate dose range, Dex can effectively attenuate the surgical stress response, provide intraoperative hemodynamic stability, and improve the patient recovery quality. High-dose Dex can delay patient awakening from anesthesia and increase the incidence of bradycardia. This randomized controlled trial aimed to investigate the effects of low-dose intravenous Dex premedication in patients undergoing laparoscopic cholecystectomy (LC).

ELIGIBILITY:
Inclusion Criteria:

* age 18-64 years with planned LC
* American Society of Anesthesiologists (ASA) physical status of Grade I or II
* body mass index (BMI) of 20-30 kg/m2 .

Exclusion Criteria:

* severe cardiovascular
* cerebrovascular disease
* severe endocrine
* liver, kidney
* neurological
* blood system disease
* preoperative respiratory infection or asthma
* history of opioid addiction
* allergy to the drugs used in this study
* psychosocial disease or cognitive dysfunction.
* incomplete case report form or lost to follow-up and failed to undergo an effectiveness and safety assessment
* LC converted to open surgery
* severe hemodynamic instability during surgery
* surgical duration >2 h .

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
the incidence of bradycardia | 24 hours
  heart rate of study patients will be recorded every 5 min during surgery and every 1 hour postoperative